CLINICAL TRIAL: NCT04018911
Title: Assessment of Novel Sound Changing Principles in Hearing Instruments to Determine Their Application
Brief Title: Assessment of Novel Sound Changing Principles in Hearing Instruments to Determine Their Application - 2019_20
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sonova AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Sonova2019_20
Record Dates: First submitted 2019-06-20; First posted 2019-07-15 (Actual); Last update posted 2019-10-11 (Actual); Status verified 2019-10

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss | interventions — Hearing Aids

STUDY DESIGN:
Intervention Model Description: Each participant will be treated with each sound changing principle (Noise Reduction principle (NR)) in a randomized order.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Hearing Aid standard NR_1 (Active Comparator): Hearing Aid with standard Noise Reduction (NR) serves as reference condition.
  Interventions: Device: Hearing Aid with standard Noise Reduction (NR_1)
- Hearing Aid with NR_2 (Experimental): NR_2: Noise Reduction principle 2
  Interventions: Device: Hearing Aid with NR_2
- Hearing Aid with NR_3 (Experimental): NR_3: Noise Reduction principle 3
  Interventions: Device: Hearing Aid with NR_3
- Hearing Aid with NR_4 (Experimental): NR_4: Noise Reduction principle 4
  Interventions: Drug: Hearing Aid with NR_4

INTERVENTIONS:
Device: Hearing Aid with standard Noise Reduction (NR_1) — Hearing Aid with standard Noise Reduction (NR) Each participant will be fitted with the 4 different Noise Reduction (Sound Changing) principles on the same hearing aid, saved to 4 manual programs (ensures exact same hearing loss compensation for each intervention). Noise Reduction principle is a sound processing algorithm to remove noise from a speech signal to improve the speech intelligibility and comfort. The active comparator condition is the state of the art Noise Reduction principle.
  Arms: Hearing Aid standard NR_1
Device: Hearing Aid with NR_2 — Each participant will be fitted with the 4 different Noise Reduction (Sound Changing) principles on the same hearing aid, saved to 4 manual programs. Noise Reduction principle is a sound processing algorithm to remove noise from a speech signal to improve the speech intelligibility and comfort. The experimental conditions (novel NR principle) vary in their parametrization to result in different degrees of noise suppression and good speech quality.
  Arms: Hearing Aid with NR_2
Device: Hearing Aid with NR_3 — Each participant will be fitted with the 4 different Noise Reduction (Sound Changing) principles on the same hearing aid, saved to 4 manual programs. Noise Reduction principle is a sound processing algorithm to remove noise from a speech signal to improve the speech intelligibility and comfort. The experimental conditions (novel NR principle) vary in their parametrization to result in different degrees of noise suppression and good speech quality.
  Arms: Hearing Aid with NR_3
Drug: Hearing Aid with NR_4 — Each participant will be fitted with the 4 different Noise Reduction (Sound Changing) principles on the same hearing aid, saved to 4 manual programs. Noise Reduction principle is a sound processing algorithm to remove noise from a speech signal to improve the speech intelligibility and comfort. This experimental condition combines standard NR and novel NR principle to result in different degrees of noise suppression and good speech quality.
  Arms: Hearing Aid with NR_4

SUMMARY:
A methodical evaluation of novel sound changing principles in CE-labelled Sonova brand hearing instruments (e.g. Phonak hearing instruments) is intended to be conducted on hearing impaired participants. These sound changing principles are enabled by respective hearing instrument technologies and hearing instrument algorithms. The aim of the study is to investigate and asses strength and weaknesses of these novel sound changing principles in terms of hearing performance to determine their application in hearing instruments (Phase of development). Both, objective laboratory measurements as well as subjective evaluations in real life environment will be carried out. This will be a controlled, single blinded and randomised active comparator clinical evaluation which will be conducted mono centric at Sonova AG Headquarter based in Stäfa

ELIGIBILITY:
Inclusion Criteria:

* Healthy outer ear (without previous surgical procedures)
* Ability to fill in a questionnaire conscientiously
* Informed Consent as documented by signature

Exclusion Criteria:

* Contraindications to the MD in this study, e.g. known hypersensitivity or allergy to the investigational product

  * Limited mobility and not in the position to attend weekly appointments
  * Limited ability to describe listening impressions/experiences and the use of the hearing aid
  * Inability to produce a reliable hearing test result
  * Massively limited dexterity
  * Known psychological problems
  * Known central hearing disorders
  * colour blinded

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-06-03 (Actual); Primary Completion 2019-08-19 (Actual); Study Completion 2019-09-16 (Actual)

PRIMARY OUTCOMES:
sound quality ratings | 4 weeks
  The sound quality ratings will be assessed with the aid of a Multi-Stimulus Test. The data, serving as the primary outcome measure, are collected in the laboratory and will use a continuous rating scale. The scale ranges from 0 "very bad" to 100 "very good" in increments of 1.

SECONDARY OUTCOMES:
Oldenburg sentence test & reaction time task | 3 weeks
  A dual task paradigm will be used in which the Oldenburg Sentence test in noise will be administered as a primary task, and the subject will press a button as fast as possible when a light appears on a screen as a secondary task. The aim is to recall as many words from the presented sentence at a predefined SNR and press the button as fast as possible at the same time. The data derived, serving as secondary outcome measure are he Signal to noise ratio (SNR) in decibel (dB) where a 50% speech reception threshold is reached and the reaction time (RT) in seconds and the number of missed stimuli. and number of false alarms missed data rate.
Oldenburg Sentence test (Olsa) | 4 weeks
  Oldenburg Sentence test in noise will be administered as single task. The aim is to recall as many words from the presented sentence at different signal to noise ratios until the 50% threshold is reached. The data derived, serving as secondary outcome measure are the Signal to noise ratio (SNR) in decibel (dB) where a 50% speech reception threshold is reached.
Adaptive Categorial Listening Effort Scaling (ACALES) | 3 weeks
  The ACALES procedure determines self-reported individual listening effort on a scale from "extreme effort" to "no effort" within a signal-to-noise ratio range that corresponds to individual subject perceptions.
  The data, serving as a secondary outcome, are a set of points on a categorial scale (subjectively perceived listening effort) as a function of different SNRs.
qualitative interview form | 3 weeks
  A qualitative questionnaire with predefined questions and comment sections to gather information on individual perceptions regarding the 3 experimental conditions to the active comparator ( see study arms/ interventions for detailed descriptions) during different laboratory-based complex acoustic scenes. The data collected from this questionnaire are scores on a continuous rating scale ranging from "0" (worst) to "10"( best).

OTHER OUTCOMES:
Non-verbal Trail Making Test A & B | 1 week
  The Trail Making Test is a neuropsychological test of visual attention and task switching. It consists of two parts in which the subject is instructed to connect a set of 25 dots as quickly as possible while still maintaining accuracy. The data, serving as an outcome measure, are time-to-complete the set in seconds.
color-word-interference test by J.R.Stroop | 1 week
  The color-word- interference test ("Farb-Wort-Interferenztest nach J.R.Stroop" (version: "Günther Bäumler")) is a neuropsychological test of visual attention and interferer suppression and will be carried out in the laboratory. In the first trial, the subject has to read the names of colours written on a card as fast and accurately as possible. In the second trial, the subject has to name the colour ink of filled boxes on a card as quickly and accurately as possible. In the third trial, the names of colours are written on a card in a dissimilarly coloured ink. The participant must read aloud the written words, whilst ignoring the colour of the ink. The data, serving as an outcome measure, are time-to-complete the sets in seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Juliane Raether, Principal Investigator — Sonova AG
Locations (1):
- Sonova AG, Stäfa, Switzerland

IPD SHARING:
Plan to Share IPD: No